CLINICAL TRIAL: NCT01727479
Title: The Effect of Ribose on Performance and Recovery in Athletes
Brief Title: Ribose and Sport Performance
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Laval University (Other)
Collaborators: Atrium Innovations (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Prevention
Other Study IDs: 2012-048; INAF-2012-048
Record Dates: First submitted 2012-11-02; First posted 2012-11-16 (Estimated); Last update posted 2016-12-05 (Estimated); Status verified 2016-12

CONDITIONS: Sports
Keywords: Peak VO2 consumption; 3km time trial; fatigue perception; lactate; time to complete
MeSH Terms: interventions — Ribose

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (2):
- Ribose (Experimental): After each of the 3km time trial (3 in total), consumption of ribose incorporated in a sports drink.
  Interventions: Other: Ribose
- Placebo (Placebo Comparator): After each of the 3km time trial (3 in total), consumption of placebo incorporated in a sports drink.
  Interventions: Other: Placebo

INTERVENTIONS:
Other: Ribose — After each of the 3km time trial (3 in total), participants will be asked to drink the experimental product (or placebo) incorporated in a sports drink.
  Arms: Ribose
Other: Placebo
  Arms: Placebo

SUMMARY:
Investigate the acute effect of ribose supplementation on performance and recovery in athletes.

ELIGIBILITY:
Inclusion Criteria:

* Men and women
* Training volume > 7hrs/week
* VO2 max > 40 and 45 mg/kg/min (for women and men respectively)
* Otherwise healthy individuals

Exclusion Criteria:

* Pregnant or breastfeeding women
* Individuals with endocrine disorders, hypercholesterolemia, cardiovascular diseases, gut diseases, cancer, anemia, hypoglycemia
* Medication for lipids, diabetes, hypertension, inflammation, autoimmune diseases, mood disorders
* Excessive alcohol consumption (more than two drinks by day for men, one for women), smoking, drug use, supplements or natural products consumption during the study

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Actual)
Dates: Start 2012-08; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

PRIMARY OUTCOMES:
Change in time to complete the third of 3 consecutive 3km time trials on bike | baseline and 1 week

SECONDARY OUTCOMES:
Performance on the 3 consecutive 3km time trials on bike | baseline and 1 week
  Performance measures: peak power (watts/kg), mean power (watts/kg), time to peak power (sec), total work (kJ) and maximum cadence (RPMmax)

OTHER OUTCOMES:
Fatigue perception after each of the 3 consecutive 3km time trials on bike | baseline and 1 week
  Post-exercise fatigue perception on visual analog scale (VAS)
Peak Vo2 consumption during each of the 3km time trials on bike | baseline and 1 week

CONTACTS AND LOCATIONS:
Overall Officials: Benoît Lamarche, PhD, Principal Investigator — Institute on nutraceuticals and functional foods
Locations (1):
- Université Laval, Québec, Quebec, Canada